CLINICAL TRIAL: NCT02463955
Title: Exploration of the Pleural Cavity Using a fleXible endoscoPe Under Two-Lung ventilatiOn With contRollEd Capnothorax
Brief Title: Exploration of the Pleural Cavity Using a fleXible endoscoPe
Acronym: EXPLORE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never start
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/182/HP; 2014-A01660-47 (Other: ANSM)
Record Dates: First submitted 2015-04-30; First posted 2015-06-04 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pleural Effusion
Keywords: flexible endoscopy
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thoracoscopy (Experimental): 1. experimental intervention (flexible video endoscope)
  2. reference procedure (video-rigid thoracoscope)
  Interventions: Device: flexible video endoscope; Device: video-rigid thoracoscope

INTERVENTIONS:
Device: flexible video endoscope — Thoracoscopy is done using flexible video endoscope
Device: video-rigid thoracoscope — Thoracoscopy is done using video-rigid thoracoscope

SUMMARY:
EXPLORE is a first-in-human study of single port transdiaphragmatic thoracoscopy using a flexible gastro-intestinal endoscope under two-lung ventilation with controlled capnothorax.

DETAILED DESCRIPTION:
Thoracoscopy is usually performed either with rigid thoracoscopes, or with flexible bronchoscopes. The latter is less invasive and less expensive, but flexible bronchoscopes are difficult to manipulate within the pleural cavity and do not provide an adequate orientation within the pleural space. It is therefore associated with a lower diagnostic yield than thoracoscopy with rigid thoracoscopes. On the other hand, rigid thoracoscopes are associated with more pain, a higher cost, and usually require one-lung ventilation. Gastro-intestinal endoscopes allow a better orientation than bronchoscopes in cavities, and have wider operative channels. The EXPLORE study investigates the feasibility and safety of single port transdiaphragmatic thoracoscopy using a flexible gastro-intestinal endoscope under two-lung ventilation with controlled capnothorax.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pleural effusion affirmed by chest radiography,
* Indication thoracoscopy, asked by the pulmonologist or thoracic surgeon for diagnostic investigation and / or pleural symphysis
* Inpatient or outpatient,
* Women of childbearing age having an effective contraceptive coverage (combined oral contraceptives or intrauterine device or tubal ligation); a negative pregnancy test should be obtained,
* For postmenopausal women, menopause confirmation of diagnosis,

Exclusion Criteria:

* Pleural effusion compression,
* Pleural effusion infected or suspected of infection,
* Febrile patient (> 38 ° C)
* Parapneumonic effusion
* Immunosuppression (eg, neutropenia <1G / L, immunosuppressive therapy, ...)
* Portage known multidrug-resistant germ or S. aureus resistant to methicillin,
* Clinical suspicion of tuberculosis,
* Patients who have already been treated by pleurodesis,
* Contraindication to general anesthesia,
* Contraindication of prophylactic antibiotics,
* Contraindication to pleurodesis agent
* Increased bleeding risk,
* No one deprived of liberty by an administrative or judicial decision or protected adult subject (under guardianship)
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Completeness of the pleural cavity exploration using the flexible endoscope | at 0 hours
  Two independent experts will visualize the video-recordings of the intervention and evaluate the completeness of the exploration using a standardized score.

SECONDARY OUTCOMES:
Outcome of a complication | at 0 hours
  Complications are defined by any of the following: any grade >2 event of the Clavien-Dindo classification, a documented or suspected infection, a non programmed admission to the hospital, a prolongation of hospitalization, or death.
Outcome of a complication | at 4 hours
  Complications are defined by any of the following: any grade >2 event of the Clavien-Dindo classification, a documented or suspected infection, a non programmed admission to the hospital, a prolongation of hospitalization, or death.
Outcome of a complication | Day 7
  Complications are defined by any of the following: any grade >2 event of the Clavien-Dindo classification, a documented or suspected infection, a non programmed admission to the hospital, a prolongation of hospitalization, or death.
Outcome of a complication | 1 month
  Complications are defined by any of the following: any grade >2 event of the Clavien-Dindo classification, a documented or suspected infection, a non programmed admission to the hospital, a prolongation of hospitalization, or death.
Results of the microbiological analysis of samples collected on the endoscope seven days before the intervention | Day -7 : 7 days before the intervention
Results of the microbiological analysis of samples collected on the endoscope the day of the intervention | at 0 hours
Completeness of the pleural cavity exploration using the standard three-ports thoracoscopy with one-lung ventilation | at 0 hours
  Two independent experts will visualize the video-recordings of the intervention and evaluate tee completeness of the exploration using a standardized score.
Diagnostic yield of biopsies performed with the flexible endoscope | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: BASTE Jean Marc, MD, Principal Investigator — University Hospital, Rouen